CLINICAL TRIAL: NCT03080935
Title: A Multicenter, Open-label, Single-arm, Extension Study to Assess Long-term Safety of Evolocumab Therapy in Subjects With Clinically Evident Cardiovascular Disease in Selected European Countries
Brief Title: Fourier Open-label Extension Study in Subjects With Clinically Evident Cardiovascular Disease in Selected European Countries
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Amgen business decision to close study early
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160250; 2016-004066-26 (EudraCT Number)
Record Dates: First submitted 2017-03-10; First posted 2017-03-15 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — evolocumab

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Evolocumab (Experimental): Single arm study administering Evolocumab.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Subjects will receive Evolocumab 140 mg every 2 weeks (Q2W) or 420 mg monthly (QM), according to the subject's preference.
  Other Names: AMG 145

SUMMARY:
This is a multicenter, open-label extension (OLE) study designed to assess the extended long-term safety of evolocumab in subjects who have completed the FOURIER trial (Study 20110118). Approximately 1600 subjects will be enrolled in this study. This study will continue for 260 weeks (approximately 5 years).

DETAILED DESCRIPTION:
This is a multicenter, open-label extension (OLE) study designed to assess the extended long-term safety of evolocumab in subjects who have completed the FOURIER trial (Study 20110118). FOURIER is a randomized placebo-controlled study of evolocumab, in patients with clinically evident atherosclerotic CVD on stable effective statin therapy. Subjects at sites participating in FOURIER OLE (Study 20160250) who are eligible and have signed the FOURIER OLE informed consent will be enrolled after completion of FOURIER.

The FOURIER OLE study requires laboratory assessments at day 1, week 12, and thereafter approximately every 6 months from day 1; the corresponding blood samples will be processed using a central laboratory.

Upon enrollment in FOURIER OLE study, subjects will receive evolocumab 140 mg every 2 weeks (Q2W) or 420 mg monthly (QM) according to their preference. Frequency and corresponding dose of administration can be changed at any scheduled time point where evolocumab is supplied to the subject, provided the appropriate supply is available. It is recommended that subjects continue the same background lipid-lowering therapy (LLT), including statin, as taken during FOURIER.

This study will continue for 260 weeks (approximately 5 years). Subjects ending administration of evolocumab should continue study assessments until the end of study. All subjects will be followed and complete procedures/assessments from enrollment through the date of study termination unless the subject has withdrawn consent, irrespective of whether the subject is continuing to receive treatment.

All deaths and cardiovascular events of interest will be reviewed by an independent external Clinical Events Committee (CEC), using standardized definitions.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures.
* Subject had completed FOURIER (Study 20110118) while still receiving assigned Investigational Product.

Exclusion Criteria:

* Permanent discontinuation of Investigational Product during FOURIER for any reason including an adverse event or serious adverse event.
* Currently receiving treatment in another investigational device or drug study, or less than 4 weeks since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Subject has known sensitivity to any of the active substances or excipients (eg, sodium acetate) to be administered during dosing.
* Females who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment with evolocumab and for an additional 15 weeks after treatment with evolocumab discontinues.
* Female subjects of childbearing potential unwilling to use an acceptable method of effective contraception during treatment and for an additional 15 weeks after the last dose of protocol-required therapies.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (85):
- Belgium (16):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Imelda Ziekenhuis vzw, Bonheiden
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Cliniques universitaires de Bruxelles Hopital Erasme, Brussels
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Medif sprl, Gozée
  - Centre Hospitalier Universitaire de Tivoli, La LouviÃ¨re
  - Centres Hospitaliers Jolimont - Hopital de Jolimont, La LouviÃ¨re
  - Centre Hospitalier Regional de la Citadelle, LiÃ¨ge
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Algemeen Ziekenhuis Turnhout, Turnhout
- Denmark (14):
  - Aalborg Hospital, Aalborg
  - Center for Clinical and Basic Research Aalborg, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Centre for Clinical and Basic Research Ballerup, Ballerup Municipality
  - Sydvestjysk Sygehus, Esbjerg
  - Frederiksberg/Bispebjerg Hospitaler, Frederiksberg
  - Glostrup Hospital, Glostrup Municipality
  - Hvidovre Hospital, Hvidovre
  - Amager Hospital, København S
  - Odense Universitetssygehus, Odense
  - Sjaellands Universitetshospital, Roskilde, Roskilde
  - Svendborg Sygehus, Svendborg
  - Center for Clinical and Basic Research Vejle, Vejle
  - Regionshospitalet Viborg, Viborg
- France (13):
  - Centre Hospitalier Regional Universitaire de Besancon, Hopital Jean Minjoz, Besançon
  - Centre Hospitalier RÃ©gional Universitaire de Tours - HÃ´pital Trousseau, Chambray-lès-Tours
  - Hopital Louis Pasteur, Le Coudray
  - Centre Hospitalier Regional Universitaire de Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Universitaire de Nantes - Hopital Guillaume et Rene Laennec, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Hopital Lariboisiere, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Centre Hospitalier de Pau - Hopital Francois Mitterrand, Pau
  - Centre Hospitalier Universitaire de Reims - Hopital Robert Debre, Reims
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
  - Centre Hospitalier Intercommunal Haute Saone, Vesoul
- Germany (17):
  - Universitaets-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Klinische Forschung Berlin GbR, Berlin
  - Vivantes Klinikum NeukÃ¶lln, Berlin
  - Deutsches Rotes Kreuz Kliniken Berlin KÃ¶penick, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Sankt-Johannes-Hospital, Dortmund
  - Gesellschaft fur Wissens und Technologietransfer der Technischen Uni Dresden, Dresden
  - Ambulantes Herzzentrum Kassel, Kassel
  - UniversitÃ¤tsklinikum KÃ¶ln, KÃ¶ln
  - Otto von Guericke UniversitÃ¤t Magdeburg, Magdeburg
  - Johannes Gutenberg UniversitÃ¤t Mainz, Mainz
  - Herz-GefÃ¤ÃŸ-Zentrum Nymphenburg am Klinikum Dritter Orden, MÃ¼nchen
  - Deutsches Herzzentrum MÃ¼nchen des Freistaates Bayern, MÃ¼nchen
  - Robert Bosch Krankenhaus, Stuttgart
  - UniversitÃ¤tsklinikum Ulm, Ulm
  - Forschungszentrum Ruhr, Witten
  - Helios UniversitÃ¤tsklinikum Wuppertal, Wuppertal
- Italy (9):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Centro Cardiologico Monzino, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Fondazione Toscana Gabriele Monasterio, Stabilimento Ospedaliero di Pisa, Pisa
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
- Portugal (6):
  - Hospital Garcia de Orta, EPE, Almada
  - Centro Hospitalar e Universitario de Coimbra EPE, Coimbra
  - Centro Hospitalar Cova da Beira, EPE - Hospital Pero da Covilha, Covilha
  - Hospital Cuf Infante Santo, Lisbon
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Sao Francisco Xavier, Lisbon
  - Centro Hospitalar de Setubal EPE Hospital de Sao Bernardo, Setúbal
- Sweden (10):
  - Falu Lasarett, Falun
  - Helsingborgs Lasarett, Helsingborg
  - LÃ¤nssjukhuset Ryhov, JÃ¶nkÃ¶ping
  - Sunderby Sjukhus, Luleå
  - Skanes Universitetssjukhus, Lund
  - Capio Citykliniken, Lund
  - Universitetssjukhuset Ã-rebro, Örebro
  - Ostersunds sjukhus, Östersund
  - Akardo MedSite, Stockholm
  - Norrlands Universitetssjukhus, Umeå

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] O'Donoghue ML, Giugliano RP, Wiviott SD, Atar D, Keech A, Kuder JF, Im K, Murphy SA, Flores-Arredondo JH, Lopez JAG, Elliott-Davey M, Wang B, Monsalvo ML, Abbasi S, Sabatine MS. Long-Term Evolocumab in Patients With Established Atherosclerotic Cardiovascular Disease. Circulation. 2022 Oct 11;146(15):1109-1119. doi: 10.1161/CIRCULATIONAHA.122.061620. Epub 2022 Aug 29. PMID 36031810
- [Background] McClintick DJ, O'Donoghue ML, De Ferrari GM, Ferreira J, Ran X, Im K, Lopez JAG, Elliott-Davey M, Wang B, Monsalvo ML, Atar D, Keech A, Giugliano RP, Sabatine MS. Long-Term Efficacy of Evolocumab in Patients With or Without Multivessel Coronary Disease. J Am Coll Cardiol. 2024 Feb 13;83(6):652-664. doi: 10.1016/j.jacc.2023.11.029. PMID 38325990
- [Derived] Katsiki N, Athyros VG, Mikhailidis DP, Mantzoros C. Proprotein convertase subtilisin-kexin type 9 (PCSK9) inhibitors: Shaping the future after the further cardiovascular outcomes research with PCSK9 inhibition in subjects with elevated risk (FOURIER) trial. Metabolism. 2017 Sep;74:43-46. doi: 10.1016/j.metabol.2017.04.007. Epub 2017 Apr 20. No abstract available. PMID 28477848
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension of study 20110118 (NCT01764633). Eligible participants were enrolled after the completion of the 20110118 study. 1600 participants were enrolled at 86 centers in Belgium, Germany, Denmark, France, Italy, Portugal, and Sweden from 13 March 2017 to 04 March 2022.
Pre-assignment Details: 1600 participants were enrolled and 1599 of those participants received study drug.
Groups:
- Placebo Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study: Participants in the parent study who received placebo subcutaneous injections either Q2W or QM, and received evolocumab 140 mg Q2W or 420 mg QM in the open label extension, according to the participant's preference.
- Evolocumab Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study: Participants in the parent study who received evolocumab either Q2W or QM, and received evolocumab 140 mg Q2W or 420 mg QM in the open label extension according to the participants preference.
Period: Overall Study
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study
Started | 745 | 855
Completed | 695 | 786
Not Completed | 50 | 69
Not completed — Death | 34 | 50
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 11 | 15

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants is made up of all of the participants that received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study | Total
Number analyzed (Participants) | 745 | 854 | 1599
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (9.1) | 62.6 (8.9) | 62.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 151 | 289
  Male | 607 | 703 | 1310
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 24 | 41
  Not Hispanic or Latino | 728 | 830 | 1558
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Black or African American | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  White | 706 | 797 | 1503
  Multiple | 0 | 0 | 0
  Other | 38 | 53 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: All adverse event summaries for the primary analysis of the primary endpoint (OLE study period only) included all treatment-emergent events reported on the Event electronic case report form (eCRF), including CEC positively reviewed events and disease-related events.
Time Frame: Up to 5 years
Population: OLE Safety Analysis Set which included all participants who received at least 1 dose of open-label evolocumab in the OLE study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study
Number analyzed (Participants) | 745 | 854
Participants | 686 | 810

2. Secondary Outcome: Percent Change of Low-density Lipoprotein Cholesterol (LDL-C) From Baseline at Each Scheduled Visit
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 72, Week 96, Week 120, Week 144, Week 168, Week 192, Week 216, Week 260
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study
Number analyzed (Participants) | 745 | 854
Percent Change
  Week 12: number analyzed (Participants) | 724 | 822
  Week 12 | -66.32 (26.88) | -67.24 (25.23)
  Week 24: number analyzed (Participants) | 726 | 837
  Week 24 | -66.48 (27.52) | -66.47 (28.11)
  Week 48: number analyzed (Participants) | 714 | 823
  Week 48 | -62.61 (26.60) | -63.45 (26.03)
  Week 72: number analyzed (Participants) | 708 | 819
  Week 72 | -65.58 (28.13) | -65.33 (28.42)
  Week 96: number analyzed (Participants) | 705 | 811
  Week 96 | -64.58 (27.01) | -63.43 (28.80)
  Week 120: number analyzed (Participants) | 695 | 797
  Week 120 | -64.26 (28.31) | -63.10 (29.56)
  Week 144: number analyzed (Participants) | 489 | 590
  Week 144 | -66.79 (29.22) | -65.13 (31.96)
  Week 168: number analyzed (Participants) | 661 | 750
  Week 168 | -65.28 (27.55) | -63.55 (29.60)
  Week 192: number analyzed (Participants) | 633 | 722
  Week 192 | -65.02 (27.93) | -62.46 (26.39)
  Week 216: number analyzed (Participants) | 653 | 741
  Week 216 | -64.92 (27.93) | -62.46 (28.32)
  Week 260: number analyzed (Participants) | 373 | 426
  Week 260 | -66.45 (29.84) | -64.72 (29.50)

3. Secondary Outcome: Percentage of Participants Who Achieved an LDL-C Level < 40 mg/dL
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 72, Week 96, Week 120, Week 144, Week 168, Week 192, Week 216, Week 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study | Evolocumab Once Every 2 Weeks (Q2W) or Once Every Month (QM) in Parent Study
Number analyzed (Participants) | 745 | 854
Percentage of Participants
  Baseline in parent study | 0 [0.0 to 0.5] | 0 [0.0 to 0.4]
  Week 12: number analyzed (Participants) | 724 | 822
  Week 12 | 72.8 [69.4 to 75.9] | 72.5 [69.4 to 75.4]
  Week 24: number analyzed (Participants) | 726 | 837
  Week 24 | 72.9 [69.5 to 76.0] | 73.4 [70.3 to 76.2]
  Week 48: number analyzed (Participants) | 714 | 823
  Week 48 | 66.5 [63.0 to 69.9] | 68.0 [64.8 to 71.1]
  Week 72: number analyzed (Participants) | 708 | 819
  Week 72 | 73.2 [69.8 to 76.3] | 72.3 [69.1 to 75.2]
  Week 96: number analyzed (Participants) | 705 | 811
  Week 96 | 71.1 [67.6 to 74.3] | 69.2 [65.9 to 72.3]
  Week 120: number analyzed (Participants) | 695 | 797
  Week 120 | 70.9 [67.5 to 74.2] | 68.6 [65.3 to 71.8]
  Week 144: number analyzed (Participants) | 489 | 590
  Week 144 | 75.3 [71.2 to 78.9] | 72.2 [68.5 to 75.7]
  Week 168: number analyzed (Participants) | 661 | 750
  Week 168 | 72.3 [68.8 to 75.6] | 69.3 [65.9 to 72.5]
  Week 192: number analyzed (Participants) | 633 | 722
  Week 192 | 71.6 [67.9 to 74.9] | 66.3 [62.8 to 69.7]
  Week 216: number analyzed (Participants) | 653 | 741
  Week 216 | 72.1 [68.6 to 75.4] | 67.3 [63.9 to 70.6]
  Week 260: number analyzed (Participants) | 373 | 426
  Week 260 | 76.1 [71.6 to 80.2] | 68.8 [64.2 to 73.0]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Placebo in Parent Study: Participants with Placebo in Parent Study
- Evolocumab in Parent Study: Participants with Evolocumab in Parent Study
Arm/Group | Placebo in Parent Study | Evolocumab in Parent Study
All-Cause Mortality (participants affected / at risk) | 35/745 | 51/855
Serious Adverse Events (participants affected / at risk) | 323/745 | 410/854
Other Adverse Events (participants affected / at risk) | 451/745 | 528/854
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo in Parent Study (N=745) | Evolocumab in Parent Study (N=854)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Necrotic lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 4 | 7
Acute myocardial infarction (Cardiac disorders) | 18 | 15
Angina pectoris (Cardiac disorders) | 26 | 24
Angina unstable (Cardiac disorders) | 15 | 13
Aortic valve calcification (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 15 | 22
Atrial flutter (Cardiac disorders) | 1 | 2
Atrioventricular block (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 3
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 17 | 27
Cardiac failure acute (Cardiac disorders) | 2 | 6
Cardiac failure chronic (Cardiac disorders) | 6 | 5
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiorenal syndrome (Cardiac disorders) | 1 | 0
Chronic coronary syndrome (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 6 | 10
Coronary artery occlusion (Cardiac disorders) | 2 | 2
Coronary artery stenosis (Cardiac disorders) | 5 | 11
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Coronary ostial stenosis (Cardiac disorders) | 0 | 1
Dressler's syndrome (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 3 | 0
Left ventricular failure (Cardiac disorders) | 0 | 2
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Low cardiac output syndrome (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 4
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 6 | 9
Myocardial ischaemia (Cardiac disorders) | 7 | 3
Palpitations (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 1 | 1
Sinoatrial block (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 2
Ventricular extrasystoles (Cardiac disorders) | 2 | 1
Ventricular fibrillation (Cardiac disorders) | 3 | 3
Ventricular tachycardia (Cardiac disorders) | 8 | 4
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Von Hippel-Lindau disease (Congenital, familial and genetic disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 3
Adrenal haemorrhage (Endocrine disorders) | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Blepharitis (Eye disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Corneal oedema (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 2
Keratopathy (Eye disorders) | 0 | 1
Lens dislocation (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 5
Colitis microscopic (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enlarged uvula (Gastrointestinal disorders) | 1 | 0
Gastric cyst (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 2
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 2
Peritoneal haematoma (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Chest discomfort (General disorders) | 1 | 2
Chest pain (General disorders) | 4 | 7
Death (General disorders) | 0 | 2
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fibrosis (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 2
Impaired healing (General disorders) | 1 | 1
Incarcerated hernia (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Necrosis (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 10
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Stent-graft endoleak (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Unevaluable event (General disorders) | 1 | 1
Vascular stent occlusion (General disorders) | 2 | 0
Vascular stent stenosis (General disorders) | 3 | 2
Vascular stent thrombosis (General disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 2
Biliary polyp (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 3
Cholecystitis acute (Hepatobiliary disorders) | 4 | 9
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 5
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess jaw (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 4
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 3
COVID-19 (Infections and infestations) | 6 | 5
COVID-19 pneumonia (Infections and infestations) | 0 | 3
Campylobacter gastroenteritis (Infections and infestations) | 2 | 4
Cellulitis (Infections and infestations) | 2 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 1
Dermo-hypodermitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 7 | 4
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 1
Herpes zoster cutaneous disseminated (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 5
Infectious pleural effusion (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1
Mediastinal abscess (Infections and infestations) | 0 | 1
Meningitis streptococcal (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 15 | 19
Pneumonia aspiration (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 3 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 2 | 2
Prostatitis Escherichia coli (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 3 | 2
Septic embolus (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 4 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Stomatococcal infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 4
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 3 | 4
Vascular device infection (Infections and infestations) | 0 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 2
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 3 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 4
Electric injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 2
Hyphaema (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Medical device monitoring error (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 1
Muscle contusion (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 3
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Restenosis (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 2
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 3
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 4
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Vascular anastomosis aneurysm (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 2
Vascular graft stenosis (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood pressure orthostatic (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Cardiac function test abnormal (Investigations) | 0 | 1
Echocardiogram abnormal (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio abnormal (Investigations) | 0 | 1
Oxygen saturation abnormal (Investigations) | 0 | 1
SARS-CoV-2 antibody test positive (Investigations) | 1 | 0
Transvalvular pressure gradient increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 2
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 5
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 1
Overweight (Metabolism and nutrition disorders) | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 1
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 6
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 | 15
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 7 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angiosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo maligna stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancoast's tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Amputation stump pain (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 2 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 6
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 2 | 0
Dementia (Nervous system disorders) | 0 | 1
Dementia with Lewy bodies (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 2 | 0
Essential tremor (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 8 | 14
Memory impairment (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 2 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Peripheral nerve lesion (Nervous system disorders) | 0 | 1
Piriformis syndrome (Nervous system disorders) | 1 | 0
Post-traumatic headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 3
Sciatic nerve neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 2 | 2
Seizure (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 10 | 10
Transient global amnesia (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 9 | 3
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Device material issue (Product Issues) | 0 | 1
Device occlusion (Product Issues) | 1 | 0
Device physical property issue (Product Issues) | 1 | 0
Device power source issue (Product Issues) | 0 | 2
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 3
Eating disorder (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 8
Calculus bladder (Renal and urinary disorders) | 1 | 1
Calculus urethral (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 4 | 5
Nephropathy (Renal and urinary disorders) | 1 | 0
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Urinoma (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 | 5
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 2
Prostatomegaly (Reproductive system and breast disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Coronary revascularisation (Surgical and medical procedures) | 0 | 1
Ileectomy (Surgical and medical procedures) | 1 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Mitral valve repair (Surgical and medical procedures) | 0 | 1
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1
Aneurysm (Vascular disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 4 | 3
Aortic stenosis (Vascular disorders) | 1 | 1
Arterial stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 2
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 4 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 3
Intermittent claudication (Vascular disorders) | 3 | 2
Ischaemic limb pain (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 12 | 12
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 2 | 2
Peripheral artery stenosis (Vascular disorders) | 4 | 4
Peripheral ischaemia (Vascular disorders) | 3 | 4
Peripheral vascular disorder (Vascular disorders) | 1 | 5
Peripheral vein stenosis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Vascular pain (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo in Parent Study (N=745) | Evolocumab in Parent Study (N=854)
Atrial fibrillation (Cardiac disorders) | 37 | 49
Cataract (Eye disorders) | 42 | 32
Chest pain (General disorders) | 40 | 29
Bronchitis (Infections and infestations) | 32 | 43
Influenza (Infections and infestations) | 37 | 53
Nasopharyngitis (Infections and infestations) | 75 | 111
Pneumonia (Infections and infestations) | 42 | 41
Diabetes mellitus (Metabolism and nutrition disorders) | 60 | 57
Arthralgia (Musculoskeletal and connective tissue disorders) | 61 | 75
Back pain (Musculoskeletal and connective tissue disorders) | 50 | 70
Myalgia (Musculoskeletal and connective tissue disorders) | 55 | 47
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 50
Dizziness (Nervous system disorders) | 33 | 43
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 40
Hypertension (Vascular disorders) | 132 | 150

LIMITATIONS AND CAVEATS:
This study was terminated to coincide with the completion of study 20130295 (NCT02867813). The study was not terminated due to any safety findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT03080935/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT03080935/SAP_001.pdf